CLINICAL TRIAL: NCT02967874
Title: Safety/Efficacy of Intra-articularly Administrated Autologous Adipose -Derived Stromal Vascular Fraction Cells in Treatment of Knee Osteoarthritis
Brief Title: Autologous Adipose-Derived Stromal Vascular Fraction Cells for Osteoarthritis Treatment
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Russian Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alexander A Ostanin, Head of Clinical Department, Russian Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFCI-10/11/2015
Record Dates: First submitted 2016-11-16; First posted 2016-11-18 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis; Joint Disease; Osteoarthritis,Knee; Arthritis, Degenerative; Osteoarthrosis; Osteoarthrosis Deformans
Keywords: Adipose -Derived Stromal Vascular Fraction Cells; Knee Osteoarthritis; Intra-articular Administration; Liposuction
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Osteoarthritis, Knee | interventions — Hyaluronic Acid

ARMS (2):
- Intra-articular auto-SVFs injection (Experimental): The participants will undergo a standard liposuction to harvest adipose tissue. The adipose tissue will then be processed to obtain the SVFs.
  This group of subjects (n=16) will receive a single injection of auto-SVFs into affected knees (3.0 mL cell suspension/joint).
  Interventions: Procedure: Intra-articular auto-SVFs injection
- Intra-articular Hyaluronic Acid (Active Comparator): This group of subjects (n=11) will receive a single injection of Synocrom Forte 2% into affected knees (1.0 mL/joint).
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Procedure: Intra-articular auto-SVFs injection — Liposuction under local anesthesia followed by single intra-articular injection of auto-SVFs under the ultrasound navigation
  Arms: Intra-articular auto-SVFs injection
Drug: Hyaluronic Acid — Single intra-articular injection of Synocrom Forte 2% under the ultrasound navigation
  Other Names: Synocrom Forte
  Arms: Intra-articular Hyaluronic Acid

SUMMARY:
Adipose-derived stromal vascular fraction cells (SVFs) include regenerative cell populations (hematopoietic cells, pericytes, endothelial cells and progenitors, stromal/stem cells) and thus are potentially important as new therapeutic tools for the repair and regeneration of acute and chronically damaged tissues.

The general objective of this study is to evaluate safety and clinical efficacy of a single intra-articular injection of freshly isolated auto-SVFs for the treatment of patients with knee osteoarthritis (OA). This study uses autologous adipose-derived SVFs, as therapeutic agent and intra-articular administration, as a mode of delivery. Expected clinical effects: a treatment reduces pain, increases function and reduces stiffness in the knees of osteoarthritic subjects.

DETAILED DESCRIPTION:
Subcutaneous human adipose tissue is an abundant and accessible cell source for applications in tissue engineering and regenerative medicine. Methods to extract stromal/stem cells from the waste products of abdominoplasty, cosmetic surgery, and liposuction are now well developed. Routinely, the adipose tissue is digested with collagenase or related enzymes to release a heterogeneous population of SVF cells. The SVF cells can be used directly or can be cultured in plastic ware to select and expand an adherent population known as adipose-derived stromal/stem cells.

Osteoarthritis is the most common joint disease that affects at least 20% of the world population. The disease usually begins at the age of 40 years. Radiographic signs of osteoarthritis are diagnosed in 50% of people aged 55 years and 80% - over 75 years. OA can cause severe pain and stiffness in the affected joints, thus reducing joint's functionality. Therefore a treatment that would reduce pain/stiffness and increase joint function would be of benefit to many people. Safety and feasibility of SVFs in OA patients have been shown in few clinical studies.

This trial is a prospective, controlled, non-randomized, non-blinded, interventional study to determine safety and efficacy of a single injection of freshly isolated autologous SVFs into the knees of osteoarthritic patients (Grade II-III). In experimental group the participants (n=16) will undergo a standard liposuction to harvest adipose tissue, then the adipose tissue will be processed to obtain the SVFs and patients will receive a single intra-articular injection of auto-SVFs into affected knees under the ultrasound navigation. In parallel control group the participants (n=11) will receive a single intra-articular injection of hyaluronic acid (Synocrom Forte 2%) under the ultrasound navigation. The safety of auto-SVFs injection will be evaluated by assessment of the frequency and nature of adverse events occurring during or immediately after the procedure, and up to the one year following treatment. Patients will be monitored during 1, 3, 6 and 12- month's visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 85 Years (Adult, Senior)
* Grade II or Grade III osteoarthritis of the knee joints using Kellgren-Lawrence grading scale (K-L Grade) as diagnosed using weight bearing X-ray and physician review, and/or MRI
* Patients must have continued pain in the knee despite conservative therapies for at least 3 months
* Patients must be able to tolerate all study procedures
* Patients must be willing to voluntarily give written Informed Consent to participate in the study before any procedures are performed
* Patients must be willing to be available for all baseline, treatment and follow-up examinations required by protocol

Exclusion Criteria:

* Subjects with a BMI > 35
* Subjects who have had an injection in either knee in the prior 4 weeks, including corticosteroids, drugs of hyaluronic acid or platelet rich plasma (PRP).
* Subjects who have had surgery of either knee within 6 months prior to the screening visit
* Subjects those are allergic to drugs for local anesthesia
* Psychiatric disorders
* Hepatic or renal dysfunctions
* Hemodynamic or respiratory instability
* HIV or uncontrolled bacterial, fungal, or viral infections
* Autoimmune diseases (rheumatoid arthritis, lupus arthropathy, psoriatic arthritis, etc)
* Pregnancy
* Malignancy
* Participation in other clinical trials

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-03; Primary Completion 2019-06 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
The number of patients with adverse events | up to 12 months after treatment
  The safety of intra-articular injection of auto-SVFs will be evaluated by assessment of the frequency and nature of adverse events during or immediately after the procedure, and up to the 12-months following treatment

SECONDARY OUTCOMES:
Change in pain score on the Visual Analogue Scale (VAS) at all follow-up visits | Baseline, 1, 3, 6 and 12 months after treatment
  The severity of joint pain, which is determined by the patient from 0 (no pain) to 10 points (unbearable pain), will be evaluated.
Change in Knee injury and Osteoarthritis Outcome Score (KOOS) at all follow-up visits | Baseline, 1, 3, 6 and 12 months after treatment
  KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Change in Ultrasonography of the knee joints | Baseline, 3, 6 and 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Elena R Chernykh, MD, PhD, Study Chair — Institute of Fundamental and Clinical Immunology; Alexander A Ostanin, MD, PhD, Principal Investigator — Institute of Fundamental and Clinical Immunology
Locations (1):
- Institute of Fundamental and Clinical Immunology, Novosibirsk, Russia

REFERENCES:
- [Background] Michalek J, Moster R, Lukac L, Proefrock K, Petrasovic M, Rybar J, Capkova M, Chaloupka A, Darinskas A, Michalek J Sr, Kristek J, Travnik J, Jabandziev P, Cibulka M, Holek M, Jurik M, Skopalik J, Kristkova Z, Dudasova Z. WITHDRAWN: Autologous adipose tissue-derived stromal vascular fraction cells application in patients with osteoarthritis. Cell Transplant. 2015 Jan 20. doi: 10.3727/096368915X686760. Online ahead of print. PMID 25706817
- [Background] Garza GR, Palomera T, Dumanian GA, Dos-Anjos S. Use of autologous adipose-derived stromal vascular fraction to treat osteoarthritis of the knee: a feasibility and safety study. J Regen Med. 4(1), 2015 doi:10.4172/2325-9620.1000119